CLINICAL TRIAL: NCT02952807
Title: Sequential Versus Concurrent Use of Vaginal Misoprostol Plus Foley Catheter for Induction of Labor
Brief Title: Vaginal Misoprostol and Foley Catheter for Induction of Labor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, IBRAHIM ABD ELGAFOR, assistant lecturer, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2016-11

CONDITIONS: Induction of Labor Affected Fetus / Newborn
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sequential (Active Comparator): sequential use of vaginal misoprotol Plus Foley Catheter for Induction of Labor.
  Interventions: Drug: Misoprostol; Device: Foley Catheter
- Concurrent (Active Comparator): Concurrent Use of Vaginal misoprostol Plus Foley Catheter for Induction of Labor.
  Interventions: Drug: Misoprostol; Device: Foley Catheter

INTERVENTIONS:
Drug: Misoprostol — vaginal Misoprostol Plus Foley Catheter
  Other Names: cytotec
Device: Foley Catheter

SUMMARY:
to compare between sequential and concurrent use of vaginal misopristol plus foleys catheter for induction of labor

DETAILED DESCRIPTION:
two groups of patients who are eligible for labor induction were randomized to either sequential use of vaginal misopristol plus foleys catheter or concurrent use of vaginal misopristol plus foleys catheter.

ELIGIBILITY:
Inclusion Criteria:

* Indication for labour induction Term pregnancy with alive fetus Bishop score less than five

Exclusion Criteria:

* Age less than 18 years Previous uterine scar Nonvertex presentation Non-reassuring fetal status Fetal anomalies Fetal growth restriction Genital bleeding Tumors, malformations and/or ulcers of vulva, perineum or vagina

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2016-01; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
induction delivery interval (time from starting induction to delivery) | 48hours
  safety issue

SECONDARY OUTCOMES:
Need of oxytocin for augmentation of labour | 48h
  safety issue
Number of doses needed to bring on labour | 48h
  safety issue
Failed induction (failure to elicit contraction after 72 hours) | 72h
  safety issue
Hyperstimulation syndrome | 24h
  safety issue
Cesarean section | 72h
  safety issue
Severe neonatal morbidity or perinatal death | 28 days
  safety issue
Serious maternal morbidity or maternal death | 42 days
  safety issue

CONTACTS AND LOCATIONS:
Overall Officials: ibrahim A el sharkwy, MD, Principal Investigator — FACULTY OF MEDICINE ,ZAGAZIG UNIVERSITY
Locations (1):
- Zagazig University, Zagazig, Egypt

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264